CLINICAL TRIAL: NCT05022992
Title: Effects of a Single Bout of Resistance Training Session on Hormonal Response in Pre-pubertal and Pubertal Boys
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Umeå University (Other)
Responsible Party: Principal Investigator, Apostolos Theos, Associate Professor, Umeå University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2020-03179
Record Dates: First submitted 2021-06-11; First posted 2021-08-26 (Actual); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: Hormones; Cytokines
MeSH Terms: interventions — Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resistance Training Session (Experimental): Resistance training. Heavy resistance training. 10 reps x 3 set of upper- and lower-body resistance exercises
  Interventions: Other: Resistance Training
- Control (No Intervention): Control activity. None-exercising. 30 min of rest

INTERVENTIONS:
Other: Resistance Training — Both groups will perform a resistance training session consisted of 10 reps x 3 set of upper- and lower-body resistance exercises.
  Arms: Resistance Training Session

SUMMARY:
: Resistance training induces strength gains in both children and adolescents. Exercise training is linked to anabolic functions through the GH-IGF-I axis. This has been demonstrated in studies showing a higher activity of GH and IGF-I in fitter adolescents and adults. Exercise also stimulates pro-inflammatory cytokines (IL-1β, IL-6, TNF-α) that suppress the GH-IGF-I axis. This has been observed in endurance-type training, while resistance training has received less attention.

Boys experience a significant physiological muscle-growth change during puberty that is associated with increases in boys androgen levels. How maturation affects the hormonal response to resistance training in boys is unclear. Therefore, the purpose of the study is to compare the acute effects of a single bout of resistance training on hormones and pro-inflammatory cytokines in pre-pubertal and pubertal boys.

DETAILED DESCRIPTION:
Preliminary measurements:

Preliminary testing will include anthropometric measurements of body mass, height, body fat percentage, and lean leg volume (LLV). The maturation stage will be determined according to the Tanner scale. There will also be an assessment of maximal strength testing to determine exercise intensity for each individual. Two familiarization sessions will be conducted for muscular strength before the muscular strength testing session.

Main trial A venous blood sample will be collected pre-exercise at resting condition. The trial will start with a standardized warm-up followed by a short (20-30 min), high-intensity whole-body resistance training session. Venous blood samples will be collected immediately after the completion of the training session and during the recovery period.

ELIGIBILITY:
Inclusion Criteria:

* Healthy boys (n=40)
* Physically active, defined as a minimum of 2 years experience in a sports club
* Biological age range: 20 pre-pubertal (Tanner I-II) - 20 pubertal (Tanner III-IV) boys
* No previous experience of structured resistance training

Exclusion Criteria:

* Chronic diseases that affect full participation
* Injuries that limit full participation

Ages: 9 Years to 17 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes
Enrollment: 40 (Estimated)
Dates: Start 2021-09 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Growth Hormone Baseline | Baseline testing before the exercise intervention (Pre values)
  Blood Concentration of Growth Hormone
Change from Baseline Growth Hormone Post exercise | Right after the completion of the exercise intervention (Post values)
  Blood Concentration of Growth Hormone
Change from Baseline Growth Hormone 15 minutes post exercise | 15 minutes after the completion of the exercise intervention (Post-15 values)
  Blood Concentration of Growth Hormone
Change from Baseline Growth Hormone 30 minutes post exercise | 30 minutes after the completion of the exercise intervention (Post-30 values)
  Blood Concentration of Growth Hormone
Insulin-like Growth Factor-1 Baseline | Baseline testing before the exercise intervention (Pre values)
  Blood concentration of Insulin-like Growth Factor-1
Change from Baseline Insulin-like Growth Factor-1 Post exercise | Right after the completion of the exercise intervention (Post values)
  Blood concentration of Insulin-like Growth Factor-1
Change from Baseline Insulin-like Growth Factor-1 15 minutes Post exercise | 15 minutes after the completion of the exercise intervention (Post-15 values)
  Blood concentration of Insulin-like Growth Factor-1
Change from Baseline Insulin-like Growth Factor-1 30 minutes Post exercise | 30 minutes after the completion of the exercise intervention (Post-30 values)
  Blood concentration of Insulin-like Growth Factor-1

SECONDARY OUTCOMES:
Cortisol Baseline | Baseline testing before the exercise intervention (Pre values)
  Blood concentration of Cortisol
Change from Baseline Cortisol Post exercise | Right after the completion of the exercise intervention (Post values)
  Blood concentration of Cortisol
Change from Baseline Cortisol 15 minutes Post exercise | 15 minutes after the completion of the exercise intervention (Post-15 values)
  Blood concentration of Cortisol
Change from Baseline Cortisol 30 minutes Post exercise | 30 minutes after the completion of the exercise intervention (Post-30 values)
  Blood concentration of Cortisol
Testosterone Baseline | Baseline testing before the exercise intervention (Pre values)
  Blood concentration of testosterone
Change from Baseline Testosterone Post Exercise | Right after the completion of the exercise intervention (Post values)
  Blood concentration of testosterone
Change from Baseline Testosterone 15 minutes Post Exercise | 15 minutes after the completion of the exercise intervention (Post-15 values)
  Blood concentration of testosterone
Change from Baseline Testosterone 30 minutes Post Exercise | 30 minutes after the completion of the exercise intervention (Post-30 values)
  Blood concentration of testosterone
Interleukin-6 Baseline | Baseline testing before the exercise intervention (Pre values)
  Blood concentration of Interleukin-6
Change from Baseline Interleukin-6 Post Exercise | Right after the completion of the exercise intervention (Post values)
  Blood concentration of Interleukin-6
Change from Baseline Interleukin-6 15 minutes Post Exercise | 15 minutes after the completion of the exercise intervention (Post-15 values)
  Blood concentration of Interleukin-6
Change from Baseline Interleukin-6 30 minutes Post Exercise | 30 minutes after the completion of the exercise intervention (Post-30 values)
  Blood concentration of Interleukin-6
Interleukin-1 alpha Baseline | Baseline testing before the exercise intervention (Pre values)
  Blood concentration of Interleukin-1 alpha
Change from Baseline Interleukin-1 alpha Post Exercise | Right after the completion of the exercise intervention (Post values)
  Blood concentration of Interleukin-1 alpha
Change from Baseline Interleukin-1 alpha 15 minutes Post Exercise | 15 minutes after the completion of the exercise intervention (Post-15 values)
  Blood concentration of Interleukin-1 alpha
Change from Baseline Interleukin-1 alpha 30 minutes Post Exercise | 30 minutes after the completion of the exercise intervention (Post-30 values)
  Blood concentration of Interleukin-1 alpha
Tumor Necrosis Factor alpha Baseline | Baseline testing before the exercise intervention (Pre values)
  Blood concentration of Tumor Necrosis Factor alpha
Change from Baseline Tumor Necrosis Factor alpha Post Exercise | Right after the completion of the exercise intervention (Post values)
  Blood concentration of Tumor Necrosis Factor alpha
Change from Baseline Tumor Necrosis Factor alpha 15 minutes Post Exercise | 15 minutes after the completion of the exercise intervention (Post-15 values)
  Blood concentration of Tumor Necrosis Factor alpha
Change from Baseline Tumor Necrosis Factor alpha 30 minutes Post Exercise | 30 minutes after the completion of the exercise intervention (Post-30 values)
  Blood concentration of Tumor Necrosis Factor alpha
Sex Hormone Binding Globulin Baseline | Baseline testing before the exercise intervention (Pre values)
  Blood concentration of Sex Hormone Binding Globulin
Change from Baseline Baseline Sex Hormone Binding Post Exercise | Right after the completion of the exercise intervention (Post values)
  Blood concentration of Sex Hormone Binding Globulin
Change from Baseline Baseline Sex Hormone Binding 15 minutes Post Exercise | 15 minutes after the completion of the exercise intervention (Post-15 values)
  Blood concentration of Sex Hormone Binding Globulin
Change from Baseline Sex Hormone Binding Globulin 30 minutes Post Exercise | 30 minutes after the completion of the exercise intervention (Post-30 values)
  Blood concentration of Sex Hormone Binding Globulin

CONTACTS AND LOCATIONS:
Overall Officials: Apostolos Theos, PhD, Principal Investigator — Umeå University
Locations (1):
- Umeå Movement and Exercise Laboratory, Umeå University, Umeå, Västerbotten County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jansson D, Lundberg E, Rullander AC, Domellof M, Lindberg AS, Andersson H, Theos A. Hormonal and inflammatory responses in prepubertal vs. pubertal male children following an acute free-weight resistance training session. Eur J Appl Physiol. 2025 Feb;125(2):381-392. doi: 10.1007/s00421-024-05603-2. Epub 2024 Sep 11. PMID 39259397